CLINICAL TRIAL: NCT04937231
Title: Comparative Effects of Aerobic Exercises, Resistance Training and Combined Training on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/00880 Mahnoor Shabbir
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Aerobic Exercises; Resistance Training; Combined Training
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercises (Experimental): Treadmill and Cycle ergometer
  Interventions: Other: Aerobic exercises
- Resistance exercises (Experimental): unilateral leg press, Bilateral leg press, unilateral arm curls
  Interventions: Other: Resistance exercises
- Combined training (Experimental): Treadmill and Cycle ergometer along with resistive Training
  Interventions: Other: Combined training

INTERVENTIONS:
Other: Aerobic exercises — For Week 1 and 2 : Treadmill 3-5days/weeks
  Intensity:
  50-70 vo2 peak Or HRR 60-80% Duration of 10-20 minutes For Week 3 and 4; Cycle ergometer 3-5days/weeks
  Intensity:
  50-70 vo2 peak Or HRR 60-80% Duration of 30-40 minutes
  Arms: Aerobic exercises
Other: Resistance exercises — For Week 1 and 2; 2 x 10 rep (unilateral leg press) 4x 12 reps (Bilateral leg press
  1 x 8 rep ( unilateral arm curls For Week 3 and 4; 1 x 10 reps Shoulder press
  1 x15 rep Bilateral knee extension
  1 x 10 reps Bilateral arm curls
  Arms: Resistance exercises
Other: Combined training — For Week 1 and 2; Aerobic exercise on Treadmill along with dumbbell to perform upper limb exercises (biceps curls, side curls extensions, upright row, back fly) and used Thera band to perform lower limb exercises for 10-20 minutes For Week 3 and 4; Aerobic exercise on Treadmill along with dumbbell and Thera band to perform upper limb and lower limb exercises for 30-40 minutes
  Arms: Combined training

SUMMARY:
To compare the effectiveness of aerobic training and resistance training and combined training on heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with ejection fraction greater than 35%

Exclusion Criteria:

* Patients with unstable angina
* Patients who had severe pain in the lower limbs
* Patients with Blood pressure greater than 190/120mmHg were excluded
* Patients who had positive contraindication for cardiac rehabilitation were not admitted in this study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 4th week
  Hospital Anxiety and Depression Scale (HADS) is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. Changes from the Baseline will be measured.
Minnesota living with heart failure questionnaire | 4th week
  Minnesota living with heart failure questionnaire (MLHFQ) is a self-administered, 21-item disease-specific instrument for patients with heart failure. MLHFQ is an instrument which has been widely used to assess quality of life among heart failure patients. Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life. The MLHFQ has two domains; physical domain (eight items, score range from 0 to 40) and emotional domain (five items, score range from 0 to 25). Changes from the Baseline will be measured
6 Min walk test (Distance in meters) | 4th Week
  Changes from the baseline, 6 Min Walk Distance (6 MWD) was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Peak VO2 with formula | 4th Week
  A generalized equation can be used to determined Peak rate of oxygen consumption (peak VO2). The generalized equation can be used to accurately estimate mean peak VO2 from mean 6 MWD, among groups of patients with diverse diseases without the need for cardiopulmonary exercise testing. The equation is:
  Mean peak VO2(ml/kg/mins) = 4.948 + 0.023*Mean 6 MWD (meter) Changes From the Baseline will be measured.
Heart Rate/Pulse Rate | 4th Week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter. Crossly it was measure by Chest belt (Polar Heart Rate monitors). Changes from the Baseline will be measure.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Rawalpindi Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No